CLINICAL TRIAL: NCT06928675
Title: CANTO - Cell-free DNA in Acute Stroke
Brief Title: Cell-free DNA in Acute Stroke
Acronym: CANTO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00235; ko24grosse2
Record Dates: First submitted 2025-03-18; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: cell-free DNA; stroke etiologies; reperfusion; secondary emboli; stroke subtypes
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cell-free DNA (cfDNA) is an important pro-inflammatory and prothrombotic mediator. With this study the investigators aim to gain new insights into the role of cfDNA in stroke and to perform a combined analysis of cfDNA in the hyperacute phase of the disease using blood and thrombus analyses. The main objectives are to analyse cfDNA in different stroke etiologies, to investigate the relationship between cfDNA and important procedural factors such as secondary embolisation and reperfusion outcomes, to analyse the correlation between blood and thrombus content of cfDNA and to investigate the specific source of cfDNA in distinct stroke subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke due to large vessel occlusion (LVO) who require mechanical thrombectomy (detected in CT-Scan or MRI-Scan)
* 18 years of age

Exclusion Criteria:

* Patients currently undergoing immunological therapies.
* Patients with immunological diseases
* Patients with systemic infections at the time of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male or female patients over 18 years of age presenting with acute ischemic stroke due to large vessel occlusion (LVO) who require mechanical thrombectomy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Stroke Etiology | at day 1
  Descriptive comparison of cell-free DNA in cerebral thrombi regarding stroke etiology

SECONDARY OUTCOMES:
Correlation cfDNA concentration and perfusion outcome | at day 1
  cfDNA abount in blood and thromi is assessed in relation to thrombectomy outcomes including perfusion outcome
Correlation cfDNA concentration and secondary embolism | at day 1
  cfDNA abount in blood and thromi is assessed in relation to thrombectomy outcomes including secondary embolism
Correlation cfDNA concentration and thrombus fragmentation. | at day 1
  cfDNA abount in blood and thromi is assessed in relation to thrombectomy outcomes including thrombus fragmentation
Measures of cfDNA as a marker of systemic inflammation | at day 1
  to correlate cfDNA amount in blood and thrombi
90-day functional outcomes | up to 3 month
  to examine the association between cfDNA concentrations in blood and thrombi with 90-day functional outcomes.
  To assess functional outcomes, the modified Rankin Scale (mRS) is evaluated via a structured telephone interview on day 90. A favorable outcome is defined as an mRS score of 0 to 2 points, while an unfavorable outcome is defined as an mRS score of 3 to 5 points.

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit Grosse, PD Dr. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland